CLINICAL TRIAL: NCT02721121
Title: Comparison of Circumferential Pulmonary Vein Isolation Alone Versus Linear Ablation in Addition to Circumferential Pulmonary Vein Isolation for Catheter Ablation in Persistent Atrial Fibrillation: Prospective Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-0029
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- circumferential pulmonary vein isolation (Active Comparator): circumferential pulmonary vein isolation
  Interventions: Procedure: circumferential pulmonary vein isolation
- Linear ablation in addiction to pulmonary vein isolation (Experimental): Linear ablation in addiction to pulmonary vein isolation
  Interventions: Procedure: Linear ablation in addiction to circumferential pulmonary vein isolation

INTERVENTIONS:
Procedure: circumferential pulmonary vein isolation
  Arms: circumferential pulmonary vein isolation
Procedure: Linear ablation in addiction to circumferential pulmonary vein isolation
  Arms: Linear ablation in addiction to pulmonary vein isolation

SUMMARY:
The purpose of this study is to compare the clinical outcomes depending on catheter ablation strategy for persistent atrial fibrillation. After randomization, investigators will conduct circumferential pulmonary vein isolation alone in a group, and additional posterior box isolation and anterior linear ablation in the other group. Investigators will compare clinical recurrence rate, complication rate, and procedure time, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent Atrial fibrillation (20~80 years)
* LA diameter <55mm
* patients possible to anticoagulation and anti arrhythmic drug

Exclusion Criteria:

* Structural cardiac disease
* Contraindication to brain perfusion CT
* Catheter ablation history for AF,
* Cardiac surgery for AF
* active internal bleeding
* Impossible to anticoagulation or antiarrhythmic drug
* valvular AF (MA> GII, Mechanical valve, Mitral valve replacement)
* Patients with severe medical disease
* Expected survival < 1year
* Severe alcoholics, drug addiction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2016-03; Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation after catheter ablation | 12 month

SECONDARY OUTCOMES:
procedure time | 1 day
procedure related complication rate | 12 month
rate of hospitalization | 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JM, Shim J, Park J, Yu HT, Kim TH, Park JK, Uhm JS, Kim JB, Joung B, Lee MH, Kim YH, Pak HN; POBI-AF Investigators. The Electrical Isolation of the Left Atrial Posterior Wall in Catheter Ablation of Persistent Atrial Fibrillation. JACC Clin Electrophysiol. 2019 Nov;5(11):1253-1261. doi: 10.1016/j.jacep.2019.08.021. Epub 2019 Oct 30. PMID 31753429